CLINICAL TRIAL: NCT00427934
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Assess the Safety and Efficacy of Maraviroc in the Treatment of Rheumatoid Arthritis in Subjects Receiving Methotrexate
Brief Title: Maraviroc in Rheumatoid Arthritis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: See Detailed Description.
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A4001056
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Results first posted 2010-02-05 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-10

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Maraviroc

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Placebo Comparator)
  Interventions: Drug: Maraviroc Placebo
- 1 (Experimental): This study was divided into two components: safety/pharmacokinetic (PK) and proof-of-concept (POC). In the safety/PK component either 150 mg or 300 mg tablets of maraviroc was administered twice a day (BID) to 16 rheumatoid arthritis subjects for 4 weeks.
  Interventions: Drug: Maraviroc

INTERVENTIONS:
Drug: Maraviroc — 300 mg (2- 150 mg tablets) are administered by mouth twice a day (BID) for 12 weeks.
  Arms: 1
Drug: Maraviroc Placebo — Placebo tablets to match active drug. Two tablets are administered by mouth twice a day (BID) for 12 weeks.
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate whether maraviroc, an investigational drug given with methotrexate (MTX) is safe and effective in the treatment of rheumatoid arthritis in adult patients.

DETAILED DESCRIPTION:
Following a planned interim analysis in the POC component on 21 August 2008 by the internal DMC (Data Monitoring Committee) of study A4001056, the trial was discontinued due to lack of efficacy. All participating investigators/country offices and monitors were notified on 22 August 2008 to cease patient enrollment. The DMC indicated that maraviroc was well tolerated in the Rheumatoid Arthritis patients and there were no safety concerns in the study. The termination date of this trial was 07 October 2008 when the last patient last visit occurred.

ELIGIBILITY:
Inclusion Criteria:

* Must be legal age of consent
* Must have active rheumatoid arthritis based upon the American College of Rheumatology (ACR) 1987 (Revised Criteria); minimum disease criteria required for entry into the efficacy component of the study
* Must meet ACR 1991 Revised Criteria for Global Functional Status in RA, Class I, II, or III
* Must be receiving methotrexate for at least 12 weeks duration and on a stable dose for 4 weeks.

Exclusion Criteria:

* Diagnosed with any other inflammatory arthritis or a secondary non-inflammatory arthritis that would interfere with disease activity assessments.
* Subject receiving prior treatment with certain medications for rheumatoid arthritis
* Tuberculosis and/or a positive tuberculin reaction
* Significant trauma or major surgery within 2 months
* History of alcohol and/or drug abuse outside of a defined period of abstinence
* History of or a finding at screening of postural hypotension
* Any condition that would affect the oral absorption of the drug
* History of cancer and in remission less than 3 years or Grade III-IV congestive heart failure
* Having an infection of human immunodeficiency virus (HIV), Hepatitis B or C or evidence of any active infection
* Abnormalities of clinical or laboratory assessments completed at the screening visit such as elevated liver enzymes, decreased hemoglobin or an abnormal ECG
* Having a positive chemokine receptor 5 (CCR5) delta 32 mutation
* Requiring the use of certain medications
* Lactating or pregnant women or subjects have reproductive potential unwilling to use an adequate method of birth control
* Chronic or recent serious or life-threatening infection; severe , progressive and/or uncontrollable renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, cardiac, neurological disease within 12 weeks of the first dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2007-02; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (36):
- United States (17):
  - Pfizer Investigational Site, Huntington Beach, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Hamden, Connecticut
  - Pfizer Investigational Site, Meriden, Connecticut
  - Pfizer Investigational Site, New Haven, Connecticut
  - Pfizer Investigational Site, Daytona Beach, Florida
  - Pfizer Investigational Site, Port Orange, Florida
  - Pfizer Investigational Site, Savannah, Georgia
  - Pfizer Investigational Site, Moline, Illinois
  - Pfizer Investigational Site, Madisonville, Kentucky
  - Pfizer Investigational Site, Kalamazoo, Michigan
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Syracuse, New York
  - Pfizer Investigational Site, Hickory, North Carolina
  - Pfizer Investigational Site, Minot, North Dakota
  - Pfizer Investigational Site, Duncansville, Pennsylvania
- Australia (3):
  - Pfizer Investigational Site, Maroochydore, Queensland
  - Pfizer Investigational Site, Woodville, South Australia
  - Pfizer Investigational Site, Hobart, Tasmania
- Germany (2):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Leipzig
- India (2):
  - Pfizer Investigational Site, Hyderabad, Andhra Pradesh
  - Pfizer Investigational Site, Bangalore, Karnataka
- Italy (2):
  - Pfizer Investigational Site, Genova
  - Pfizer Investigational Site, Pavia
- Pfizer Investigational Site, Guadalajara, Jalisco, Mexico
- Portugal (2):
  - Pfizer Investigational Site, Coimbra
  - Pfizer Investigational Site, Lisbon
- Spain (4):
  - Pfizer Investigational Site, Santiago de Compostela, A Coruña
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Seville, Sevilla
- Ukraine (3):
  - Pfizer Investigational Site, Dnipropetrovsk
  - Pfizer Investigational Site, Kharkiv
  - Pfizer Investigational Site, Simferopol

REFERENCES:
- [Derived] Fleishaker DL, Garcia Meijide JA, Petrov A, Kohen MD, Wang X, Menon S, Stock TC, Mebus CA, Goodrich JM, Mayer HB, Zeiher BG. Maraviroc, a chemokine receptor-5 antagonist, fails to demonstrate efficacy in the treatment of patients with rheumatoid arthritis in a randomized, double-blind placebo-controlled trial. Arthritis Res Ther. 2012 Jan 17;14(1):R11. doi: 10.1186/ar3685. PMID 22251436
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4001056&StudyName=Maraviroc%20in%20Rheumatoid%20Arthritis

RESULTS

PARTICIPANT FLOW:
Groups:
- Maraviroc 150 mg BID (Pharmacokinetic [PK]): 150 mg tablet was administered by mouth twice a day (BID) for 4 weeks with stable weekly doses of methotrexate (MTX).
- Maraviroc 300 mg BID (PK): 300 mg (Two 150 mg tablets) were administered by mouth BID for 4 weeks with stable weekly doses of MTX.
- Maraviroc 300 mg BID (Proof-of-Concept [POC]): 300 mg (Two 150 mg tablets) were administered by mouth BID for 12 weeks with stable weekly doses of MTX.
- Placebo (POC): Placebo tablets to match active drug. Two tablets were administered by mouth BID for 12 weeks with stable weekly doses of MTX.
Period: Overall Study
Arm/Group | Maraviroc 150 mg BID (Pharmacokinetic [PK]) | Maraviroc 300 mg BID (PK) | Maraviroc 300 mg BID (Proof-of-Concept [POC]) | Placebo (POC)
Started | 8 | 8 | 78 | 34
Treated | 8 | 8 | 77 | 33
Completed | 7 | 8 | 55 | 19
Not Completed | 1 | 0 | 23 | 15
Not completed — Adverse Event | 1 | 0 | 5 | 4
Not completed — Lack of Efficacy | 0 | 0 | 5 | 2
Not completed — Randomized But Did Not Receive Treatment | 0 | 0 | 1 | 1
Not completed — Other | 0 | 0 | 11 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Maraviroc 150 mg BID (PK): 150 mg tablet was administered by mouth BID for 4 weeks with stable weekly doses of MTX.
- Maraviroc 300 mg BID (POC): 300 mg (Two 150 mg tablets) were administered by mouth BID for 12 weeks with stable weekly doses of MTX.
- Total: Total of all reporting groups
Arm/Group | Maraviroc 150 mg BID (PK) | Maraviroc 300 mg BID (PK) | Maraviroc 300 mg BID (POC) | Placebo (POC) | Total
Number analyzed (Participants) | 8 | 8 | 77 | 33 | 126
Age, Customized [Number; unit: Participants]
  < 18 years | 0 | 0 | 0 | 0 | 0
  18 to 44 years | 1 | 0 | 15 | 6 | 22
  45 to 64 years | 4 | 8 | 48 | 21 | 81
  > = 65 years | 3 | 0 | 14 | 6 | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 71 | 22 | 102
  Male | 4 | 3 | 6 | 11 | 24

OUTCOME MEASURES:

1. Secondary Outcome: ACR 20% Responders at Weeks 1, 2, 4, and 8
Description: A subject was an ACR 20 responder if: the counts for both tender and swollen joints had reduced by 20% or more from baseline; and 3 out of the following 5 assessments showed reduction of 20% or more from baseline assessment: Patient's Assessment of Arthritis Pain, Patient's Global Assessment of Arthritis, Physician's Global Assessment of Arthritis, HAQ-DI, and CRP. The Week 16 visit (follow-up) was designed for safety rather than efficacy, thus Week 16 ACR 20% data were collected, but not analyzed.
Time Frame: Weeks 1, 2, 4, and 8
Population: FAS. Missing values were imputed by the method of LOCF.
Measure: Number; unit: Participants
Arm/Group | Maraviroc 300 mg BID (POC) | Placebo (POC)
Number analyzed (Participants) | 77 | 33
Participants
  Week 1 | 8 | 4
  Week 2 | 12 | 5
  Week 4 | 21 | 8
  Week 8 | 23 | 7
Statistical Analysis 1: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 1; Test type: Superiority or Other; p = 0.790, Barnard/Pearson chi-square test; Percentage Difference = -1.73, 90% CI [-15.13 to 8.68] — Percentage Difference = maraviroc responders divided by the number of maraviroc participants analyzed minus placebo responders divided by the number of placebo participants analyzed
Statistical Analysis 2: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 2; Test type: Superiority or Other; p = 0.477, Barnard/Pearson chi-square test; Percentage Difference = 0.43, 90% CI [-13.67 to 11.64] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 4; Test type: Superiority or Other; p = 0.370, Barnard/Pearson chi-square test; Percentage Difference = 3.03, 90% CI [-12.85 to 16.77] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 8; Test type: Superiority or Other; p = 0.175, Barnard/Pearson chi-square test; Percentage Difference = 8.66, 90% CI [-7.07 to 22.03] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: ACR 50% Responders at Weeks 1, 2, 4, 8, and 12
Description: A subject was an ACR 50 responder if: the counts for both tender and swollen joints had reduced by 50% or more from baseline; and 3 out of the following 5 assessments showed reduction of 50% or more from baseline assessment: Patient's Assessment of Arthritis Pain, Patient's Global Assessment of Arthritis, Physician's Global Assessment of Arthritis, HAQ-DI, and CRP. The Week 16 visit (follow-up) was designed for safety rather than efficacy, thus Week 16 ACR 50% data were collected, but not analyzed.
Time Frame: Weeks 1, 2, 4, 8, and 12
Population: FAS. Missing values were imputed by the method of LOCF.
Measure: Number; unit: Participants
Arm/Group | Maraviroc 300 mg BID (POC) | Placebo (POC)
Number analyzed (Participants) | 77 | 33
Participants
  Week 1 | 1 | 0
  Week 2 | 2 | 0
  Week 4 | 2 | 2
  Week 8 | 6 | 3
  Week 12 | 8 | 3
Statistical Analysis 1: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 1; Test type: Superiority or Other; p = 0.420, Barnard/Pearson chi-square test; Percentage Difference = 1.30, 90% CI [-6.34 to 6.01] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 2; Test type: Superiority or Other; p = 0.258, Barnard/Pearson chi-square test; Percentage Difference = 2.60, 90% CI [-5.08 to 7.95] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 4; Test type: Superiority or Other; p = 1.000, Barnard/Pearson chi-square test; Percentage Difference = -3.46, 90% CI [-14.39 to 3.42] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 8; Test type: Superiority or Other; p = 0.899, Barnard/Pearson chi-square test; Percentage Difference = -1.30, 90% CI [-13.56 to 7.92] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 12; Test type: Superiority or Other; p = 0.489, Barnard/Pearson chi-square test; Percentage Difference = 1.30, 90% CI [-11.24 to 10.96] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: ACR 70% Responders at Weeks 1, 2, 4, 8, and 12
Description: A subject was an ACR 70 responder if: the counts for both tender and swollen joints had reduced by 70% or more from baseline; and 3 out of the following 5 assessments showed reduction of 70% or more from baseline assessment: Patient's Assessment of Arthritis Pain, Patient's Global Assessment of Arthritis, Physician's Global Assessment of Arthritis, HAQ-DI, and CRP. The Week 16 visit (follow-up) was designed for safety rather than efficacy, thus Week 16 ACR 70% data were collected, but not analyzed.
Time Frame: Weeks 1, 2, 4, 8, and 12
Population: FAS. Missing values were imputed by the method of LOCF.
Measure: Number; unit: Participants
Arm/Group | Maraviroc 300 mg BID (POC) | Placebo (POC)
Number analyzed (Participants) | 77 | 33
Participants
  Week 1 | 0 | 0
  Week 2 | 0 | 0
  Week 4 | 0 | 1
  Week 8 | 2 | 0
  Week 12 | 0 | 1
Statistical Analysis 1: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 4; Test type: Superiority or Other; p = 1.000, Barnard/Pearson chi-square test; Percentage Difference = -3.03, 90% CI [-13.59 to 1.28] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 8; Test type: Superiority or Other; p = 0.258, Barnard/Pearson chi-square test; Percentage Difference = 2.60, 90% CI [-5.08 to 7.95] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 12; Test type: Superiority or Other; p = 1.000, Barnard/Pearson chi-square test; Percentage Difference = -3.03, 90% CI [-13.59 to 1.28] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Change From Baseline in Tender/Painful Joint Count at Weeks 1, 2, 4, 8, and 12
Description: Change from baseline at each visit was analyzed for tender/painful joint count. Twenty-eight tender and swollen joint scores included the same joints: shoulders, elbows, wrists, metacarpophalangeal joints (MCP), proximal interphalangeal joints (PIP), and the knees. The Week 16 visit (follow-up) was designed for safety rather than efficacy, thus Week 16 tender/painful joint count data were collected, but not analyzed.
Time Frame: Baseline, Weeks 1, 2, 4, 8, and 12
Population: FAS. Missing values were imputed by the method of LOCF.
Measure: Least Squares Mean (Standard Error); unit: joint count
Arm/Group | Maraviroc 300 mg BID (POC) | Placebo (POC)
Number analyzed (Participants) | 77 | 33
joint count
  Week 1 | -0.81 (0.68) | -1.91 (0.96)
  Week 2 | -2.08 (0.76) | -2.38 (1.08)
  Week 4 | -4.00 (0.84) | -4.01 (1.20)
  Week 8 | -4.85 (0.85) | -3.24 (1.21)
  Week 12 | -4.89 (0.84) | -3.41 (1.19)
Statistical Analysis 1: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 1; Test type: Superiority or Other; p = 0.335, ANCOVA — This analysis was carried out using analysis of covariance (ANCOVA) with baseline tender/painful joint count as the covariate, treatment, region as fixed effects; Mean Difference (Final Values) = 1.10, 90% CI [-0.79 to 2.99]
Statistical Analysis 2: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 2; Test type: Superiority or Other; p = 0.816, ANCOVA — This analysis was carried out using ANCOVA with baseline tender/painful joint count as the covariate, treatment, region as fixed effects; Mean Difference (Final Values) = 0.30, 90% CI [-1.82 to 2.41]
Statistical Analysis 3: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 4; Test type: Superiority or Other; p = 0.996, ANCOVA — [p-value comment as in outcome 4, analysis 2]; Median Difference (Final Values) = 0.01, 90% CI [-2.35 to 2.36]
Statistical Analysis 4: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 8; Test type: Superiority or Other; p = 0.263, ANCOVA — [p-value comment as in outcome 4, analysis 2]; Mean Difference (Final Values) = -1.61, 90% CI [-3.98 to 0.76]
Statistical Analysis 5: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 12; Test type: Superiority or Other; p = 0.294, ANCOVA — [p-value comment as in outcome 4, analysis 2]; Mean Difference (Final Values) = -1.48, 90% CI [-3.82 to 0.85]

5. Secondary Outcome: Change From Baseline in Swollen Joint Count at Weeks 1, 2, 4, 8, and 12
Description: Change from baseline at each visit was analyzed for swollen joint count. Twenty-eight tender and swollen joint scores included the same joints: shoulders, elbows, wrists, MCP joints, PIP joints, and the knees. The Week 16 visit (follow-up) was designed for safety rather than efficacy, thus Week 16 swollen joint count data were collected, but not analyzed.
Time Frame: Baseline, Weeks 1, 2, 4, 8, and 12
Population: FAS. Missing values were imputed by the method of LOCF.
Measure: Least Squares Mean (Standard Error); unit: joint count
Arm/Group | Maraviroc 300 mg BID (POC) | Placebo (POC)
Number analyzed (Participants) | 77 | 33
joint count
  Week 1 | -1.39 (0.49) | -1.07 (0.70)
  Week 2 | -2.25 (0.61) | -2.51 (0.87)
  Week 4 | -3.93 (0.54) | -4.08 (0.77)
  Week 8 | -4.48 (0.62) | -3.03 (0.88)
  Week 12 | -3.48 (0.66) | -3.43 (0.95)
Statistical Analysis 1: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 1; Test type: Superiority or Other; p = 0.700, ANCOVA — This analysis was carried out using ANCOVA baseline swollen joint count as the covariate, treatment, region as fixed effects; Mean Difference (Final Values) = -0.32, 90% CI [-1.70 to 1.06]
Statistical Analysis 2: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 2; Test type: Superiority or Other; p = 0.799, ANCOVA — [p-value comment as in outcome 5, analysis 1]; Mean Difference (Final Values) = 0.26, 90% CI [-1.45 to 1.97]
Statistical Analysis 3: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 4; Test type: Superiority or Other; p = 0.867, ANCOVA — [p-value comment as in outcome 5, analysis 1]; Mean Difference (Final Values) = 0.15, 90% CI [-1.35 to 1.66]
Statistical Analysis 4: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 8; Test type: Superiority or Other; p = 0.167, ANCOVA — [p-value comment as in outcome 5, analysis 1]; Mean Difference (Final Values) = -1.45, 90% CI [-3.17 to 0.28]
Statistical Analysis 5: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 12; Test type: Superiority or Other; p = 0.966, ANCOVA — [p-value comment as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.05, 90% CI [-1.91 to 1.81]

6. Secondary Outcome: Change From Baseline in Patient's Assessment of Arthritis Pain at Weeks 1, 2, 4, 8, and 12
Description: The severity of arthritis was scored by the subject between 0 (no pain) and 100 (most severe pain) on a 100 mm VAS. Change from baseline at each visit was analyzed for Patient's Assessment of Arthritis Pain. The Week 16 visit (follow-up) was designed for safety rather than efficacy, thus Week 16 Patient's Assessment of Arthritis Pain data were collected, but not analyzed.
Time Frame: Baseline, Weeks 1, 2, 4, 8, and 12
Population: FAS. Missing values were imputed by the method of LOCF.
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Maraviroc 300 mg BID (POC) | Placebo (POC)
Number analyzed (Participants) | 77 | 33
scores on scale
  Week 1 | -3.96 (2.18) | -3.62 (3.10)
  Week 2 | -8.46 (2.65) | -3.20 (3.77)
  Week 4 | -8.35 (2.70) | -9.08 (3.85)
  Week 8 | -10.30 (2.98) | -8.67 (4.24)
  Week 12 | -8.30 (2.85) | -6.09 (4.06)
Statistical Analysis 1: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 1; Test type: Superiority or Other; p = 0.925, ANCOVA — This analysis was carried out using ANCOVA with baseline patient's assessment of arthritis pain as the covariate, treatment, region as fixed effects; Mean Difference (Final Values) = -0.34, 90% CI [-6.41 to 5.72]
Statistical Analysis 2: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 2; Test type: Superiority or Other; p = 0.239, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = -5.26, 90% CI [-12.62 to 2.11]
Statistical Analysis 3: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 4; Test type: Superiority or Other; p = 0.872, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.73, 90% CI [-6.79 to 8.25]
Statistical Analysis 4: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 8; Test type: Superiority or Other; p = 0.745, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = -1.63, 90% CI [-9.91 to 6.65]
Statistical Analysis 5: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 12; Test type: Superiority or Other; p = 0.644, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = -2.22, 90% CI [-10.14 to 5.71]

7. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Arthritis Pain at Weeks 1, 2, 4, 8, and 12
Description: Subjects answered: "Considering all the ways your arthritis affects you, how are you feeling today?" Subjects responded by using a 0 - 100 mm VAS where 0=very well and 100=very poorly. Change from baseline at each visit was analyzed for Patient's Global Assessment. The Week 16 visit (follow-up) was designed for safety rather than efficacy, thus Week 16 Patient's Global Assessment of Arthritis Pain data were collected, but not analyzed.
Time Frame: Baseline, Weeks 1, 2, 4, 8, and 12
Population: FAS. Missing values were imputed by the method of LOCF.
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Maraviroc 300 mg BID (POC) | Placebo (POC)
Number analyzed (Participants) | 76 | 33
scores on scale
  Week 1 | -4.70 (2.22) | -2.34 (3.13)
  Week 2 | -8.85 (2.48) | -4.88 (3.49)
  Week 4 | -10.00 (2.74) | -9.02 (3.86)
  Week 8 | -11.12 (2.93) | -3.44 (4.13)
  Week 12 | -8.55 (2.88) | -6.78 (4.06)
Statistical Analysis 1: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 1; Test type: Superiority or Other; p = 0.524, ANCOVA — This analysis was carried out using ANCOVA with baseline Patient's Global Assessment of Arthritis as the covariate, treatment, region as fixed effects; Mean Difference (Final Values) = -2.36, 90% CI [-8.49 to 3.77]
Statistical Analysis 2: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 2; Test type: Superiority or Other; p = 0.338, ANCOVA — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Final Values) = -3.96, 90% CI [-10.80 to 2.87]
Statistical Analysis 3: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 4; Test type: Superiority or Other; p = 0.830, ANCOVA — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Final Values) = -0.98, 90% CI [-8.55 to 6.58]
Statistical Analysis 4: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 8; Test type: Superiority or Other; p = 0.118, ANCOVA — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Final Values) = -7.68, 90% CI [-15.76 to 0.40]
Statistical Analysis 5: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 12; Test type: Superiority or Other; p = 0.712, ANCOVA — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Final Values) = -1.78, 90% CI [-9.73 to 6.18]

8. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Arthritis Pain at Weeks 1, 2, 4, 8, and 12
Description: Physician's evaluation based on subject's disease signs, functional capacity and physical exam. Response recorded using 5-point scale: 1=Very Good, 2=Good, 3=Fair, 4=Poor and 5=Very Poor. Change from baseline at each visit was analyzed for Physician's Global Assessment. The Week 16 visit (follow-up) was designed for safety rather than efficacy thus Week 16 Physician's Global Assessment of Arthritis Pain data were collected but not analyzed.
Time Frame: Baseline, Weeks 1, 2, 4, 8, and 12
Population: FAS. Missing values were imputed by the method of LOCF.
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Maraviroc 300 mg BID (POC) | Placebo (POC)
Number analyzed (Participants) | 75 | 32
scores on scale
  Week 1 | -0.30 (0.08) | -0.22 (0.11)
  Week 2 | -0.44 (0.09) | -0.39 (0.12)
  Week 4 | -0.49 (0.10) | -0.44 (0.13)
  Week 8 | -0.63 (0.10) | -0.37 (0.14)
  Week 12 | -0.49 (0.11) | -0.36 (0.15)
Statistical Analysis 1: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 1; Test type: Superiority or Other; p = 0.540, ANCOVA — This analysis was carried out using ANCOVA with baseline Physician's Global Assessment of Arthritis as the covariate, treatment, region as fixed effects; Mean Difference (Final Values) = -0.08, 90% CI [-0.28 to 0.13]
Statistical Analysis 2: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 2; Test type: Superiority or Other; p = 0.757, ANCOVA — [p-value comment as in outcome 8, analysis 1]; Mean Difference (Final Values) = -0.04, 90% CI [-0.28 to 0.19]
Statistical Analysis 3: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 4; Test type: Superiority or Other; p = 0.767, ANCOVA — [p-value comment as in outcome 8, analysis 1]; Mean Difference (Final Values) = -0.05, 90% CI [-0.31 to 0.21]
Statistical Analysis 4: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 8; Test type: Superiority or Other; p = 0.112, ANCOVA — [p-value comment as in outcome 8, analysis 1]; Mean Difference (Final Values) = -0.26, 90% CI [-0.52 to 0.01]
Statistical Analysis 5: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 12; Test type: Superiority or Other; p = 0.490, ANCOVA — [p-value comment as in outcome 8, analysis 1]; Mean Difference (Final Values) = -0.13, 90% CI [-0.42 to 0.17]

9. Secondary Outcome: Change From Baseline in HAQ-DI at Weeks 1, 2, 4, 8, and 12
Description: HAQ-DI assesses degree of difficulty experienced in daily activity categories (dressing/grooming, arising, eating, walking, hygiene, reach, grip and other activities) over the past week. There are 20 questions and difficulty is scored from 0 (none), 1 (some), 2 (much) and 3 (unable to do). Scores were then averaged to give the disability index (scale of 0 to 3). Change from baseline at each visit was analyzed. The Week 16 visit (follow-up) was designed for safety rather than efficacy, thus Week 16 HAQ-DI data were collected but not analyzed.
Time Frame: Baseline, Weeks 1, 2, 4, 8, and 12
Population: FAS.
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Maraviroc 300 mg BID (POC) | Placebo (POC)
Number analyzed (Participants) | 77 | 31
scores on scale
  Week 1 | -0.08 (0.05) | -0.03 (0.07)
  Week 2 | -0.22 (0.06) | -0.04 (0.08)
  Week 4 | -0.24 (0.06) | -0.18 (0.09)
  Week 8 | -0.25 (0.07) | -0.03 (0.10)
  Week 12 | -0.18 (0.08) | -0.06 (0.13)
Statistical Analysis 1: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 1; Test type: Superiority or Other; p = 0.464, ANCOVA — This analysis was carried out using ANCOVA with HAQ-DI as the covariate, treatment, region as fixed effects; Mean Difference (Final Values) = -0.06, 90% CI [-0.19 to 0.07]
Statistical Analysis 2: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 2; Test type: Superiority or Other; p = 0.068, ANCOVA — This analysis was carried out using ANCOVA with HAQ-DI as the covariate, treatment, region as fixed effects; Mean Difference (Final Values) = -0.18, 90% CI [-0.35 to -0.02]
Statistical Analysis 3: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 4; Test type: Superiority or Other; p = 0.532, ANCOVA — This analysis was carried out using ANCOVA with HAQ-DI as the covariate, treatment, region as fixed effects; Mean Difference (Final Values) = -0.06, 90% CI [-0.23 to 0.11]
Statistical Analysis 4: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 8; Test type: Superiority or Other; p = 0.063, ANCOVA — This analysis was carried out using ANCOVA with HAQ-DI as the covariate, treatment, region as fixed effects; Mean Difference (Final Values) = -0.22, 90% CI [-0.41 to -0.03]
Statistical Analysis 5: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 12; Test type: Superiority or Other; p = 0.396, ANCOVA — This analysis was carried out using ANCOVA with HAQ-DI as the covariate, treatment, region as fixed effects; Mean Difference (Final Values) = -0.12, 90% CI [-0.36 to 0.12]

10. Secondary Outcome: Change From Baseline in CRP at Weeks 1, 2, 4, 8, and 12
Description: Change from baseline at each visit were analyzed for CRP. The Week 16 visit (follow-up) was designed for safety rather than efficacy, thus Week 16 CRP data were collected, but not analyzed.
Time Frame: Baseline, Weeks 1, 2, 4, 8, and 12
Population: FAS. Missing values were imputed by the method of LOCF.
Measure: Least Squares Mean (Standard Error); unit: mg/L
Arm/Group | Maraviroc 300 mg BID (POC) | Placebo (POC)
Number analyzed (Participants) | 73 | 31
mg/L
  Week 1 | 1.20 (1.87) | 3.40 (2.67)
  Week 2 | 3.14 (2.06) | 1.81 (2.93)
  Week 4 | 3.36 (2.34) | -1.30 (3.33)
  Week 8 | 2.33 (2.10) | -1.14 (2.98)
  Week 12 | 2.35 (2.26) | 1.93 (3.22)
Statistical Analysis 1: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 1; Test type: Superiority or Other; p = 0.481, ANCOVA — This analysis was carried out using ANCOVA with CRP as the covariate, treatment, region as fixed effects; Mean Difference (Final Values) = -2.20, 90% CI [-7.36 to 2.96]
Statistical Analysis 2: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 2; Test type: Superiority or Other; p = 0.698, ANCOVA — This analysis was carried out using ANCOVA with CRP as the covariate, treatment, region as fixed effects; Mean Difference (Final Values) = 1.33, 90% CI [-4.34 to 6.99]
Statistical Analysis 3: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 4; Test type: Superiority or Other; p = 0.233, ANCOVA — This analysis was carried out using ANCOVA with CRP as the covariate, treatment, region as fixed effects; Mean Difference (Final Values) = 4.65, 90% CI [-1.79 to 11.10]
Statistical Analysis 4: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 8; Test type: Superiority or Other; p = 0.320, ANCOVA — This analysis was carried out using ANCOVA with CRP as the covariate, treatment, region as fixed effects; Mean Difference (Final Values) = 3.48, 90% CI [-2.29 to 9.25]
Statistical Analysis 5: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 12; Test type: Superiority or Other; p = 0.912, ANCOVA — This analysis was carried out using ANCOVA with CRP as the covariate, treatment, region as fixed effects; Mean Difference (Final Values) = 0.41, 90% CI [-5.81 to 6.64]

11. Secondary Outcome: Change From Baseline in Disease Activity Score Using CRP (DAS28-4[CRP]) at Weeks 1, 2, 4, 8, and 12
Description: DAS28-4 (CRP) was calculated using the following formula:
  DAS28- 4(CRP) = 0.56 √28 Tender Joint Count + 0.28 √28 Swollen Joint Count + 0.36*natural logarithm(CRP + 1) + 0.014*Patient Global Assessment + 0.96. DAS28 provides a number on a scale (0 to 10) indicating current disease activity. A score above 5.1 means high disease activity and a score below 3.2 indicates low disease activity. Change from baseline at each visit was analyzed for DAS28-4 (CRP). The Week 16 visit (follow-up) was designed for safety rather than efficacy, thus Week 16 DAS28-4 (CRP) data were collected, but not analyzed.
Time Frame: Baseline, Weeks 1, 2, 4, 8, and 12
Population: FAS. Missing values were imputed by the method of LOCF.
Measure: Least Squares Mean (Standard Error); unit: mg/L
Arm/Group | Maraviroc 300 mg BID (POC) | Placebo (POC)
Number analyzed (Participants) | 72 | 31
mg/L
  Week 1 | -0.23 (0.09) | -0.17 (0.13)
  Week 2 | -0.41 (0.12) | -0.33 (0.17)
  Week 4 | -0.64 (0.14) | -0.65 (0.19)
  Week 8 | -0.82 (0.15) | -0.51 (0.21)
  Week 12 | -0.73 (0.16) | -0.63 (0.22)
Statistical Analysis 1: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 1; Test type: Superiority or Other; p = 0.653, ANCOVA — This analysis was carried out using ANCOVA with baseline DAS28-4 (CRP) as the covariate, treatment, country as fixed effects; Mean Difference (Final Values) = -0.07, 90% CI [-0.31 to 0.18]
Statistical Analysis 2: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 2; Test type: Superiority or Other; p = 0.703, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -0.08, 90% CI [-0.41 to 0.26]
Statistical Analysis 3: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 4; Test type: Superiority or Other; p = 0.968, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = 0.01, 90% CI [-0.37 to 0.39]
Statistical Analysis 4: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 8; Test type: Superiority or Other; p = 0.210, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -0.31, 90% CI [-0.72 to 0.10]
Statistical Analysis 5: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 12; Test type: Superiority or Other; p = 0.696, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -0.10, 90% CI [-0.53 to 0.33]

12. Secondary Outcome: Change From Baseline in Mean Orthostatic Blood Pressure (BP)
Description: Supine BP was recorded after 5 minutes lying down; subjects then sat for 2 minutes then stood for 2 minutes and standing BP was recorded. Orthostatic BP = either a systolic BP drop > 20 mmHg, or diastolic BP drop > 10 mmHg and/or drop in systolic BP < 90 mmHg. If a subject met the orthostatic criteria, they were required to complete 2 additional readings to provide a triplicate reading. The means of replicate BP values were used in the analysis. Baseline = the latest non-missing value from a range of pre-treatment visits. Change from baseline to Week 16 was analyzed for orthostatic BP.
Time Frame: Baseline, 16 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Maraviroc 150 mg BID (PK) | Maraviroc 300 mg BID (PK) | Maraviroc 300 mg BID (POC) | Placebo (POC)
Number analyzed (Participants) | 8 | 8 | 77 | 33
mmHg
  Standing Systolic BP | 20.9 (13.18) | 18.0 (7.71) | 17.8 (11.25) | 17.5 (12.36)
  Supine Systolic BP | 20.9 (13.58) | 18.3 (9.51) | 17.5 (13.86) | 18.0 (11.12)
  Standing Diastolic BP | 13.0 (4.97) | 8.3 (5.65) | 11.7 (6.98) | 11.5 (5.15)
  Supine Diastolic BP | 10.3 (7.94) | 10.9 (5.08) | 12.2 (8.14) | 10.8 (5.12)

13. Primary Outcome: American College of Rheumatology (ACR) 20% Responders at Week 12
Description: A subject was an ACR 20 responder if: the counts for both tender and swollen joints had reduced by 20% or more from baseline; and 3 out of the following 5 assessments showed reduction of 20% or more from baseline assessment: Patient's Assessment of Arthritis Pain (Visual Analogue Scale [VAS]), Patient's Global Assessment of Arthritis (VAS), Physician's Global Assessment of Arthritis (Categorical), Health Assessment Questionnaire - Disability Index (HAQ-DI), and C-Reactive Protein (CRP).
Time Frame: Week 12
Population: Full Analysis Set (FAS) was defined as an intent-to-treat analysis set that included all subjects randomized to treatment who had taken at least 1 dose of study medication. Missing values were imputed by the method of last observation carried forward (LOCF).
Measure: Number; unit: Participants
Arm/Group | Maraviroc 300 mg BID (POC) | Placebo (POC)
Number analyzed (Participants) | 77 | 33
Participants | 21 | 6
Statistical Analysis 1: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Test type: Superiority or Other; p = 0.155, Barnard/Pearson chi-square test — p-value (one-sided) was based on Barnard exact test if more than 20% of expected cell counts were < 5 otherwise Pearson chi-square test; Percentage Difference = 9.09, 90% CI [-6.16 to 21.83] — [estimate comment as in outcome 1, analysis 1]

14. Secondary Outcome: Change From Baseline in Mean Heart Rate
Description: Heart rate = standing and supine at the same time the orthostatic BP measurements were obtained. Baseline was defined to be the latest non-missing value from a range of pre-treatment visits. Means of replicate values were not used.
Time Frame: Baseline, 16 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Maraviroc 150 mg BID (PK) | Maraviroc 300 mg BID (PK) | Maraviroc 300 mg BID (POC) | Placebo (POC)
Number analyzed (Participants) | 8 | 8 | 77 | 33
beats per minute (bpm)
  Standing Heart Rate | 14.6 (6.73) | 8.1 (3.64) | 11.8 (6.91) | 11.4 (8.13)
  Supine Heart Rate | 15.0 (8.28) | 10.4 (4.56) | 11.6 (6.06) | 9.2 (6.16)

15. Secondary Outcome: Number of Subjects With Categorical Absolute Vital Signs and Vital Sign Changes Compared to Baseline
Description: Baseline was defined to be the latest non-missing value from a range of pre-treatment visits. Maximum increase from baseline in supine and standing systolic BP was > = 30 mmHg, and maximum increase from baseline in supine and standing diastolic BP was > = 20 mmHg.
Time Frame: Baseline, 16 weeks
Population: FAS
Measure: Number; unit: Participants
Arm/Group | Maraviroc 150 mg BID (PK) | Maraviroc 300 mg BID (PK) | Maraviroc 300 mg BID (POC) | Placebo (POC)
Number analyzed (Participants) | 8 | 8 | 77 | 33
Participants
  Maximum Increase in Supine Systolic BP | 2 | 1 | 4 | 3
  Maximum Increase in Standing Systolic BP | 1 | 1 | 2 | 2
  Maximum Increase in Supine Diastolic BP | 1 | 1 | 8 | 0
  Maximum Increase in Standing Diastolic BP | 0 | 0 | 3 | 2

16. Secondary Outcome: Change From Baseline in 12-Lead Electrocardiogram (ECG) Parameters (RR Interval, PR Interval, QRS Complex, QT Interval, Corrected QT [QTc] Interval, QTcB Interval [Bazett's Correction], QTcF Interval [Fridericia's Correction]).
Description: Baseline was defined to be the latest non-missing value from a range of pre-treatment visits. Means of replicate values were used. QTc interval was not measured for the PK populations.
Time Frame: Baseline, 16 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Maraviroc 150 mg BID (PK) | Maraviroc 300 mg BID (PK) | Maraviroc 300 mg BID (POC) | Placebo (POC)
Number analyzed (Participants) | 8 | 8 | 77 | 33
msec
  RR Interval | 137.0 (79.18) | 114.3 (63.38) | 140.0 (70.81) | 117.6 (48.26)
  PR Interval | 19.7 (7.13) | 13.0 (6.93) | 16.2 (8.00) | 15.4 (10.47)
  QRS Complex | 7.6 (4.75) | 7.3 (4.89) | 11.3 (6.56) | 10.2 (5.35)
  QT Interval | 35.0 (19.47) | 22.5 (10.67) | 31.9 (18.74) | 28.7 (13.97)
  QTc Interval | 0 (0) | 0 (0) | 19.6 (17.69) | 20.3 (12.75)
  QTcB Interval | 23.1 (19.70) | 23.3 (9.55) | 27.9 (18.47) | 30.2 (23.88)
  QTcF Interval | 22.9 (19.64) | 17.3 (7.16) | 28.3 (18.77) | 29.8 (22.20)

17. Secondary Outcome: Change From Baseline in 12-Lead Electrocardiogram (ECG) Parameters (Heart Rate).
Description: Baseline was defined to be the latest non-missing value from a range of pre-treatment visits. Means of replicate values were used.
Time Frame: Baseline, 16 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Maraviroc 150 mg BID (PK) | Maraviroc 300 mg BID (PK) | Maraviroc 300 mg BID (POC) | Placebo (POC)
Number analyzed (Participants) | 8 | 8 | 77 | 33
bpm | 11.2 (5.82) | 8.8 (5.76) | 12.0 (6.40) | 10.5 (4.91)

18. Secondary Outcome: Number of Subjects With Categorical Absolute ECG Parameters and ECG Changes Compared to Baseline
Description: Maximum QTcB, QTcF, and QTc intervals were defined as 450 to < 480 msec, 480 to < 500 msec, or > = 500 msec.
Time Frame: Baseline, 16 weeks
Population: FAS
Measure: Number; unit: Participants
Arm/Group | Maraviroc 150 mg BID (PK) | Maraviroc 300 mg BID (PK) | Maraviroc 300 mg BID (POC) | Placebo (POC)
Number analyzed (Participants) | 8 | 8 | 77 | 33
Participants
  Maximum QTc Interval 450 to < 480 msec | 0 | 0 | 2 | 2
  Maximum QTc Interval 480 to < 500 msec | 0 | 0 | 0 | 0
  Maximum QTc Interval > = 500 msec | 0 | 0 | 0 | 0
  Maximum QTcB Interval 450 to < 480 msec | 1 | 3 | 13 | 8
  Maximum QTcB Interval 480 to < 500 msec | 0 | 0 | 2 | 1
  Maximum QTcB Interval > = 500 msec | 0 | 0 | 0 | 1
  Maximum QTcF Interval 450 to < 480 msec | 0 | 2 | 9 | 5
  Maximum QTcF Interval 480 to < 500 msec | 0 | 0 | 0 | 0
  Maximum QTcF Interval > = 500 msec | 0 | 0 | 0 | 0

19. Secondary Outcome: Change From Baseline in Short Form-36 (SF-36) Physical Component Summary at Weeks 4 and 12
Description: The SF-36 v.2 (Acute version) is a 36-item generic health status measure that measures 8 general health concepts: Physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. Each domain of the eight domains and the summary concept (physical component score) are scored to yield values between 0 (worst) and 100 (best). Change from baseline at Weeks 4 and 12 were analyzed for SF-36. Due to the termination of the study, SF-36 results for the PK component group were not analyzed.
Time Frame: Baseline, Weeks 4 and 12
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Maraviroc 300 mg BID (POC) | Placebo (POC)
Number analyzed (Participants) | 69 | 30
scores on a scale
  Week 4 | 4.33 (0.89) | 3.76 (1.25)
  Week 12 | 3.14 (1.04) | 4.81 (1.65)
Statistical Analysis 1: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 4; Test type: Superiority or Other; p = 0.698, ANCOVA — This analysis was carried out ANCOVA with baseline SF-36 score as the covariate, treatment, region as fixed effects; Mean Difference (Final Values) = 0.57, 90% CI [-1.87 to 3.01]
Statistical Analysis 2: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 12; Test type: Superiority or Other; p = 0.344, ANCOVA — This analysis was carried out ANCOVA with baseline SF-36 score as the covariate, treatment, region as fixed effects; Mean Difference (Final Values) = -1.68, 90% CI [-4.62 to 1.26]

20. Secondary Outcome: Change From Baseline in SF-36 Mental Component Summary at Weeks 4 and 12
Description: The SF-36 v.2 (Acute version) [12] is a 36-item generic health status measure that measures 8 general health concepts: Physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. Each domain of the eight domains and the summary concept (mental component score) are scored to yield values between 0 (worst) and 100 (best). Change from baseline at Weeks 4 and 12 were analyzed for SF-36. Due to the termination of the study, SF-36 results for the PK component group were not analyzed.
Time Frame: Baseline, Weeks 4 and 12
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Maraviroc 300 mg BID (POC) | Placebo (POC)
Number analyzed (Participants) | 69 | 30
scores on a scale
  Week 4 | 1.42 (1.25) | 0.72 (1.75)
  Week 12 | 1.17 (1.41) | 0.61 (2.25)
Statistical Analysis 1: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 4; Test type: Superiority or Other; p = 0.734, ANCOVA — This analysis was carried out ANCOVA with baseline SF-36 score as the covariate, treatment, region as fixed effects; Mean Difference (Final Values) = 0.70, 90% CI [-2.71 to 4.11]
Statistical Analysis 2: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Week 12; Test type: Superiority or Other; p = 0.818, ANCOVA — This analysis was carried out ANCOVA with baseline SF-36 score as the covariate, treatment, region as fixed effects; Mean Difference (Final Values) = 0.56, 90% CI [-3.50 to 4.62]

21. Secondary Outcome: Number of Subjects With Withdrawal From Study Due to Lack of Efficacy
Description: Withdrawal is the total number of withdrawals from the study. Withdrawal due to lack of efficacy was collected based on the investigator's judgement.
Time Frame: 16 weeks
Population: FAS
Measure: Number; unit: participants
Arm/Group | Maraviroc 300 mg BID (POC) | Placebo (POC)
Number analyzed (Participants) | 77 | 33
participants
  Overall Withdrawal | 22 | 14
  Withdrawal due to Lack of Efficacy | 5 | 2
Statistical Analysis 1: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Test type: Superiority or Other; p = 0.649, Fisher Exact

22. Secondary Outcome: Survival Analysis of Time to Withdrawal: Proportion of Subjects Who Did Not Withdraw From the Study Due to Lack of Efficacy.
Description: Withdrawal due to lack of efficacy was collected based on the investigator's judgement. Time to withdrawal was measured by the probability that a subject did not withdraw due to lack of efficacy by a particular visit. This was a statistical estimate (Kaplan-Meier Survival Analysis) of the probability that a participant would not withdraw due to lack of efficacy.
Time Frame: Weeks 1 to 12
Population: FAS
Measure: Number; unit: proportion
Arm/Group | Maraviroc 300 mg BID (POC) | Placebo (POC)
Number analyzed (Participants) | 77 | 33
proportion
  Week 1 (n=77, 33) | 1.00 | 1.00
  Week 2 (n=77, 32) | 1.00 | 1.00
  Week 4 (n=76, 32) | 1.00 | 1.00
  Week 8 (n=69, 31) | 0.99 | 1.00
  Week 12 (n=58, 21) | 0.93 | 0.92
Statistical Analysis 1: Comparison: Maraviroc 300 mg BID (POC) vs Placebo (POC); Test type: Superiority or Other; p = 0.9826, Log Rank

23. Secondary Outcome: Area Under the Plasma Concentration-Time Profile From Time Zero to Four Hours Postdose (AUC 0-4) for MTX at Screening and Week 1 and Maraviroc at Week 1
Description: Effect of maraviroc on the PK of MTX (comparison of AUC0-4 of MTX at screening versus at Week 1 after coadministration with 150 mg or 300 mg of maraviroc). PK was assessed at screening (MTX) and at Week 1 (maraviroc and MTX).
Time Frame: Screening (1, 2, 3, and 4 hours post-dose), Week 1 (0.5, 1, 2, 3, and 4 hours post-dose)
Population: All available PK data from the Safety/PK Component were included.
Measure: Geometric Mean (Standard Deviation); unit: ng.hr/mL
Arm/Group | Maraviroc 150 mg BID (PK) | Maraviroc 300 mg BID (PK)
Number analyzed (Participants) | 8 | 8
ng.hr/mL
  Plasma MTX (Screening) | 909.4 (422.37) | 888.9 (249.51)
  Plasma MTX (Week 1) | 1045.6 (329.93) | 844.8 (273.92)
  Plasma Maraviroc (Week 1) | 451.6 (247.33) | 1106.8 (1029.60)

24. Secondary Outcome: Maximum Observed Concentration (Cmax) During the Dosing Interval for MTX at Screening and Week 1 and Maraviroc at Week 1
Description: Effect of maraviroc on the PK of MTX (comparison of Cmax of MTX at screening versus at Week 1 after coadministration with 150 mg or 300 mg of maraviroc). PK was assessed at screening (MTX) and at Week 1 (maraviroc and MTX).
Time Frame: Screening (1, 2, 3, and 4 hours post-dose), Week 1 (0.5, 1, 2, 3, and 4 hours post-dose)
Population: All available PK data from the Safety/PK Component were included.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Maraviroc 150 mg BID (PK) | Maraviroc 300 mg BID (PK)
Number analyzed (Participants) | 8 | 8
ng/mL
  Plasma MTX (Screening) | 338.7 (143.94) | 352.1 (115.72)
  Plasma MTX (Week 1) | 403.8 (97.46) | 322.8 (104.20)
  Plasma Maraviroc (Week 1) | 199.59 (115.603) | 461.03 (365.715)

25. Secondary Outcome: Time for Cmax (Tmax) for MTX at Screening and Week 1 and Maraviroc at Week 1
Description: PK was assessed at screening (MTX) and at Week 1 (maraviroc and MTX).
Time Frame: Screening (1, 2, 3, and 4 hours post-dose), Week 1 (0.5, 1, 2, 3, and 4 hours post-dose)
Population: All available PK data from the Safety/PK Component were included.
Measure: Median (Full Range); unit: hr
Arm/Group | Maraviroc 150 mg BID (PK) | Maraviroc 300 mg BID (PK)
Number analyzed (Participants) | 8 | 8
hr
  Plasma MTX (Screening) | 2.000 [1.00 to 3.00] | 1.000 [1.00 to 3.00]
  Plasma MTX (Week 1) | 1.000 [0.50 to 2.00] | 1.500 [0.50 to 2.00]
  Plasma Maraviroc (Week 1) | 2.000 [0.50 to 3.00] | 2.500 [1.00 to 4.00]

ADVERSE EVENTS:
Arm/Group | Maraviroc 150 mg BID (PK) | Maraviroc 300 mg BID (PK) | Maraviroc 300 mg BID (POC) | Placebo (POC)
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/77 | 0/33
Other Adverse Events (participants affected / at risk) | 4/8 | 4/8 | 39/77 | 21/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Maraviroc 150 mg BID (PK) (N=8) | Maraviroc 300 mg BID (PK) (N=8) | Maraviroc 300 mg BID (POC) (N=77) | Placebo (POC) (N=33)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Goitre (Endocrine disorders) | 0 | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 1 | 1
Diplopia (Eye disorders) | 0 | 0 | 1 | 0
Glaucoma (Eye disorders) | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 1 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 6 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 4 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 2 | 1
Fatigue (General disorders) | 1 | 0 | 3 | 0
Feeling cold (General disorders) | 0 | 0 | 1 | 0
Irritability (General disorders) | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 2
Pyrexia (General disorders) | 0 | 0 | 2 | 0
Ulcer (General disorders) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 2
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 3 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 8
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 1
Headache (Nervous system disorders) | 0 | 0 | 2 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0
Hallucination, olfactory (Psychiatric disorders) | 0 | 0 | 0 | 1
Mood swings (Psychiatric disorders) | 0 | 0 | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 2 | 0
Abnormal faeces (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 0 | 0
Back injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.